CLINICAL TRIAL: NCT01548404
Title: A Randomized, Double-Blind, Placebo-Controlled, Repeat-Dose Study of the Efficacy, Safety, Tolerability, and Pharmacodynamics of Subcutaneously-Administered REGN668 in Adult Patients With Extrinsic Moderate-to-Severe Atopic Dermatitis
Brief Title: Study of Dupilumab in Adult Patients With Extrinsic Moderate-to-Severe Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R668-AD-1117
Record Dates: First submitted 2012-03-05; First posted 2012-03-08 (Estimated); Results first posted 2018-08-10 (Actual); Last update posted 2018-08-10 (Actual); Status verified 2017-11

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — dupilumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo (for Dupilumab) once weekly for 12 weeks by subcutaneous (SC) injection.
  Interventions: Drug: Placebo
- Dupilumab 300 mg (Experimental): Dupilumab 300 mg once weekly for 12 weeks by SC injection.
  Interventions: Drug: Dupilumab

INTERVENTIONS:
Drug: Placebo — Subcutaneous injection altered between back of arms, abdomen and upper thighs.
  Arms: Placebo
Drug: Dupilumab — Subcutaneous injection altered between back of arms, abdomen and upper thighs.
  Other Names: REGN668/SAR231893; Dupixent
  Arms: Dupilumab 300 mg

SUMMARY:
The primary objective was to assess the clinical efficacy of repeated subcutaneous (SC) doses of Dupilumab in adult participants with moderate-to-severe atopic dermatitis (AD).

ELIGIBILITY:
Inclusion Criteria:

The inclusion criteria included, but were not limited to the following:

1. Male or female, 18 years or older;
2. Chronic Atopic Dermatitis (AD) for at least 3 years;
3. History of inadequate response to a stable (>/= 1 month) regimen of topical corticosteroids or calcineurin inhibitors as treatment for AD within 3 months before the screening visit.

Exclusion Criteria:

1. Prior treatment with REGN668;
2. Presence of certain laboratory abnormalities at the screening visit;
3. Treatment with an investigational drug within 8 weeks ;
4. Treatment with a live (attenuated) vaccine within 12 weeks before the baseline visit;
5. Certain treatments and medical procedures, undertaken within a particular time-frame prior to the baseline visit, preclude eligibility for participation in the study;
6. Known history of human immunodeficiency virus (HIV) infection;
7. History of malignancy within 5 years before the baseline visit, with certain exceptions;
8. Planned surgical procedure during the length of the patient's participation in this study;
9. History of clinical parasite infection;
10. Any medical or psychiatric condition which in the opinion of the investigator or the sponsor's medical monitor, would place the participant at risk, interfere with participation in the study, or interfere with the interpretation of study results;
11. Pregnant or breast-feeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2012-04; Primary Completion 2013-03 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (21):
- Czechia (3):
  - Náchod
  - Svitavy
  - Ústí nad Labem
- France (3):
  - Nice
  - Pierre-Bénite
  - Toulouse
- Germany (7):
  - Berlin
  - Bonn
  - Frankfurt
  - Gera
  - Heidelberg
  - Kiel
  - Münster
- Hungary (4):
  - Kaposvár
  - Szeged
  - Szekszárd
  - Szolnok
- Poland (4):
  - Gdansk
  - Lodz
  - Lublin
  - Warsaw

REFERENCES:
- [Result] Beck LA, Thaci D, Hamilton JD, Graham NM, Bieber T, Rocklin R, Ming JE, Ren H, Kao R, Simpson E, Ardeleanu M, Weinstein SP, Pirozzi G, Guttman-Yassky E, Suarez-Farinas M, Hager MD, Stahl N, Yancopoulos GD, Radin AR. Dupilumab treatment in adults with moderate-to-severe atopic dermatitis. N Engl J Med. 2014 Jul 10;371(2):130-9. doi: 10.1056/NEJMoa1314768. PMID 25006719
- [Derived] Tsianakas A, Luger TA, Radin A. Dupilumab treatment improves quality of life in adult patients with moderate-to-severe atopic dermatitis: results from a randomized, placebo-controlled clinical trial. Br J Dermatol. 2018 Feb;178(2):406-414. doi: 10.1111/bjd.15905. Epub 2018 Jan 11. PMID 28845523

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 25 sites in Europe between 3 April 2012 and 25 June 2013. A total of 153 participants were screened in the study.
Pre-assignment Details: Out of 153 participants, 109 were randomized and treated in the study. Participants were randomized in 1:1 ratio to receive either Dupilumab 300 mg or placebo.
Period: Overall Study
Arm/Group | Placebo | Dupilumab 300 mg
Started | 54 | 55
Completed | 24 | 41
Not Completed | 30 | 14
Not completed — Adverse Event | 3 | 1
Not completed — Physician Decision | 2 | 1
Not completed — Inadequate response to study treatment | 23 | 7
Not completed — Lost to Follow-up | 2 | 0
Not completed — Withdrawal by Subject | 0 | 3
Not completed — Other than specified above | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Placebo (for Dupilumab) once weekly for 12 weeks by SC injection.
- Total: Total of all reporting groups
Arm/Group | Placebo | Dupilumab 300 mg | Total
Number analyzed (Participants) | 54 | 55 | 109
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.4 (12.29) | 33.7 (10.41) | 36.5 (11.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 24 | 51
  Male | 27 | 31 | 58
Eczema Area and Severity Index (EASI) Score [Mean (Standard Deviation); unit: units on a scale] — The EASI score is used to measure the severity and extent of atopic dermatitis (AD) and measures erythema, infiltration, excoriation and lichenification on 4 anatomic regions of the body: head, trunk, upper and lower extremities. The total EASI score ranges from 0 (minimum) to 72 (maximum) points, with the higher scores reflecting the worse severity of AD.
  units on a scale | 30.8 (13.63) | 28.4 (13.57) | 29.6 (13.59)
Investigator's Global Assessment (IGA) Score [Mean (Standard Deviation); unit: units on a scale] — IGA is an assessment scale used to determine severity of AD and clinical response to treatment on a 5-point scale (0 = clear; 1 = almost clear; 2 = mild; 3 = moderate; 4 = severe) based on erythema and papulation/infiltration. Therapeutic response was an IGA score of 0 (clear) or 1 (almost clear).
  units on a scale | 4.0 (0.69) | 3.9 (0.67) | 3.9 (0.68)
Scoring Atopic Dermatitis (SCORAD) Score [Mean (Standard Deviation); unit: units on a scale] — SCORAD is a clinical tool for assessing the severity of atopic dermatitis developed by the European Task Force on Atopic Dermatitis (Severity scoring of atopic dermatitis: the SCORAD index). Consensus Report of the European Task Force on Atopic Dermatitis. Dermatology (Basel) 186 (1): 23-31. 1993. Extent and intensity of eczema as well as subjective signs (insomnia, etc.) are assessed and scored. Total score ranges from 0 (absent disease) to 103 (severe disease).
  units on a scale | 69.1 (13.38) | 66.7 (13.82) | 67.9 (13.59)
Body Surface Area (BSA) [Mean (Standard Deviation); unit: percentage of BSA] — Body surface area affected by AD was assessed for each section of the body (the possible highest score for each region was: head and neck [9%], anterior trunk [18%], back [18%], upper limbs [18%], lower limbs [36%], and genitals [1%]). It was reported as a percentage of all major body sections combined.
  percentage of BSA | 50.8 (24.13) | 46.8 (24.55) | 48.8 (24.32)
5-D Pruritus Scale [Mean (Standard Deviation); unit: units on a scale] — The 5-D Pruritus Scale is a 1-page, 5-question tool used in clinical trials to assess 5 dimensions of background itch: degree, duration, direction, disability, and distribution. Each question corresponds to 1 of the 5 dimensions of itch; participants were to rate their symptoms over the preceding 2-week period on a 1 to 5 scale, with 5 being the most affected. After the summation of individual score, the total score ranges from 5 (least affected) to 25 (most affected).
  units on a scale | 18.7 (3.50) | 18.4 (3.04) | 18.5 (3.26)
Pruritus Numerical Rating Scale (NRS) Score [Mean (Standard Deviation); unit: units on a scale] — Pruritus NRS scale is an assessment tool that is used to report the intensity of participant's pruritus (itch), both maximum and average intensity, during a 24-hour recall period. Participants were asked the following question: how would a participant rate his itch at the worst moment during the previous 24 hours (for maximum itch intensity on a scale of 0 - 10 [0= no itch; 10= worst itch imaginable]).
  units on a scale | 5.8 (1.93) | 6.1 (1.34) | 5.9 (1.66)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Eczema Area and Severity Index (EASI) Score at Week 12- Last Observation Carried Forward (LOCF)
Description: The EASI score was used to measure the severity and extent of AD and measured erythema, infiltration, excoriation and lichenification on 4 anatomic regions of the body: head, trunk, upper and lower extremities. The total EASI score ranges from 0 (minimum) to 72 (maximum) points, with the higher scores reflecting the worse severity of AD. The efficacy data were set to be missing after use of rescue medication and after early termination visit for participants who prematurely discontinued study treatment. All missing values were imputed by LOCF.
Time Frame: Baseline to Week 12
Population: Full analysis set (FAS) population included all randomized participants who received at least one dose of study drug and had at least 1 post-baseline efficacy assessment.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | Dupilumab 300 mg
Number analyzed (Participants) | 54 | 55
percent change | -23.3 (49.26) | -74.0 (26.94)

2. Secondary Outcome: Percentage of Participants With Investigator's Global Assessment (IGA) Score of "0" or "1" at Week 12- LOCF
Description: IGA is an assessment scale used to determine severity of AD and clinical response to treatment on a 5-point scale (0 = clear; 1 = almost clear; 2 = mild; 3 = moderate; 4 = severe) based on erythema and papulation/infiltration. Therapeutic response is an IGA score of 0 (clear) or 1 (almost clear). The efficacy data were set to be missing after use of rescue medication and after early termination visit for participants who prematurely discontinued study treatment. All missing values were imputed by LOCF.
Time Frame: Week 12
Population: FAS population.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Dupilumab 300 mg
Number analyzed (Participants) | 54 | 55
percentage of participants | 7.4 | 40.0

3. Secondary Outcome: Percentage of Participants Who Achieved at Least a 50% Reduction From Baseline in the EASI Score (EASI-50) at Week 12- LOCF
Description: The EASI score was used to measure the severity and extent of AD and measured erythema, infiltration, excoriation and lichenification on 4 anatomic regions of the body: head, trunk, upper and lower extremities. The total EASI score ranges from 0 (minimum) to 72 (maximum) points, with the higher scores reflecting the worse severity of AD. EASI-50 responders were the participants who achieved ≥50% overall improvement in EASI score from baseline to Week 12. The efficacy data were set to be missing after use of rescue medication and after early termination visit for participants who prematurely discontinued study treatment. All missing values were imputed by LOCF.
Time Frame: Week 12
Population: FAS population.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Dupilumab 300 mg
Number analyzed (Participants) | 54 | 55
Percentage of participants | 35.2 | 85.5

4. Secondary Outcome: Change From Baseline in EASI Score at Week 12- LOCF
Description: as for outcome 1
Time Frame: Baseline to Week 12
Population: FAS population.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Dupilumab 300 mg
Number analyzed (Participants) | 54 | 55
Units on a scale | -6.4 (14.85) | -19.9 (11.52)

5. Secondary Outcome: Percent Change From Baseline in IGA Score at Week 12- LOCF
Description: as for outcome 2
Time Frame: Baseline to Week 12
Population: FAS population.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Placebo | Dupilumab 300 mg
Number analyzed (Participants) | 54 | 55
Percent change | -14.7 (27.37) | -49.5 (25.94)

6. Secondary Outcome: Change From Baseline in Percent Body Surface Area (BSA) Affected by Atopic Dermatitis (AD) at Week 12 - LOCF
Description: BSA affected by AD was assessed for each section of the body (the possible highest score for each region was: head and neck [9%], anterior trunk [18%], back [18%], upper limbs [18%], lower limbs [36%], and genitals [1%]). It was reported as a percentage of all major body sections combined. The efficacy data were set to be missing after use of rescue medication and after early termination visit for participants who prematurely discontinued study treatment. All missing values were imputed by LOCF.
Time Frame: Baseline to Week 12
Population: FAS population.
Measure: Mean (Standard Deviation); unit: Percentage of BSA
Arm/Group | Placebo | Dupilumab 300 mg
Number analyzed (Participants) | 54 | 55
Percentage of BSA | -9.0 (21.07) | -27.4 (22.81)

7. Secondary Outcome: Change From Baseline in Scoring Atopic Dermatitis (SCORAD) Score at Week 12- LOCF
Description: SCORAD is a clinical tool for assessing the severity of AD developed by the European Task Force on Atopic Dermatitis (Severity scoring of atopic dermatitis: the SCORAD index). Consensus Report of the European Task Force on Atopic Dermatitis. Dermatology (Basel) 186 (1): 23-31. 1993. Extent and intensity of eczema as well as subjective signs (insomnia, etc.) are assessed and scored. Total score ranges from 0 (absent disease) to 103 (severe disease). The efficacy data were set to be missing after use of rescue medication and after early termination visit for participants who prematurely discontinued study treatment. All missing values were imputed by LOCF.
Time Frame: Baseline to Week 12
Population: FAS population.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Dupilumab 300 mg
Number analyzed (Participants) | 54 | 55
Units on a scale | -9.8 (20.53) | -35.0 (19.43)

8. Secondary Outcome: Change From Baseline in Pruritus Numerical Rating Scale (NRS) to Week 12- LOCF
Description: Pruritus NRS was an assessment tool that was used to report the intensity of a participant's pruritus (itch), both maximum and average intensity, during a 24-hour recall period. Participants were asked the following question: how would a participant rate his itch at the worst moment during the previous 24 hours (for maximum itch intensity on a scale of 0 - 10 [0 = no itch; 10 = worst itch imaginable]). The efficacy data were set to be missing after use of rescue medication and after early termination visit for participants who prematurely discontinued study treatment. All missing values were imputed by LOCF.
Time Frame: Baseline to Week 12
Population: FAS population. Number of participants analyzed = participants with available data for this endpoint.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Dupilumab 300 mg
Number analyzed (Participants) | 52 | 54
units on a scale | -0.9 (2.07) | -3.5 (2.00)

9. Secondary Outcome: Change From Baseline in 5-D Pruritus Scale at Week 12
Description: The 5-D Pruritus Scale is a 1-page, 5-question tool used in clinical trials to assess 5 dimensions of background itch: degree, duration, direction, disability, and distribution. Each question corresponds to 1 of the 5 dimensions of itch; participants were to rate their symptoms over the preceding 2-week period on a 1 to 5 scale, with 5 being the most affected. After the summation of individual score, the total score ranges from 5 (least affected) to 25 (most affected).
Time Frame: Baseline to Week 12
Population: FAS population.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Dupilumab 300 mg
Number analyzed (Participants) | 54 | 55
units on a scale | -1.9 (4.28) | -7.4 (4.33)

ADVERSE EVENTS:
Time Frame: All Adverse Events (AE) were collected from signature of the informed consent form up to the final visit (Day 197) regardless of seriousness or relationship to investigational product.
Description: Reported adverse events (AEs) are treatment-emergent adverse events that is AEs that developed/worsened during the 'on treatment period' (time from first dose of study drug through the end of study (Day 197).
Arm/Group | Placebo | Dupilumab 300 mg
Serious Adverse Events (participants affected / at risk) | 7/54 | 1/55
Other Adverse Events (participants affected / at risk) | 31/54 | 38/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=54) | Dupilumab 300 mg (N=55)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Eczema herpeticum (Infections and infestations) | 1 (1) | 0 (0)
Skin bacterial infection (Infections and infestations) | 1 (1) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 4 (5) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=54) | Dupilumab 300 mg (N=55)
Eosinophilia (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 4 (4) | 0 (0)
Conjunctivitis allergic (Eye disorders) | 0 (0) | 5 (5)
Nausea (Gastrointestinal disorders) | 4 (7) | 1 (1)
Fatigue (General disorders) | 4 (5) | 5 (7)
Injection site erythema (General disorders) | 1 (1) | 4 (7)
Injection site induration (General disorders) | 3 (3) | 5 (6)
Injection site reaction (General disorders) | 1 (1) | 3 (6)
Conjunctivitis (Infections and infestations) | 2 (2) | 8 (11)
Impetigo (Infections and infestations) | 3 (3) | 1 (1)
Nasopharyngitis (Infections and infestations) | 10 (15) | 22 (33)
Oral herpes (Infections and infestations) | 0 (0) | 3 (4)
Rhinitis (Infections and infestations) | 2 (3) | 3 (3)
Neutrophil count increased (Investigations) | 3 (4) | 0 (0)
White blood cell count increased (Investigations) | 3 (4) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Headache (Nervous system disorders) | 7 (11) | 9 (12)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (4)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Not less than 45 days prior to submission for publication or presentation, the Institution shall, or cause the Principal Investigator to, provide the Sponsor with a copy of the Manuscript. The Institution shall consider in good faith any comments from the Sponsor regarding the content, and shall delete Confidential Information upon written request of the Sponsor. At the Sponsor's request, the Institution shall delay publication for an additional 60 days to allow patent applications to be filed.